CLINICAL TRIAL: NCT00406991
Title: Retinal Blood Flow and Microthrombi in Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Schepens Eye Research Institute (Other)
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2002-015; 2003P-000224; EY014812
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2006-03

CONDITIONS: Diabetes; Diabetic Retinopathy
Keywords: retinal blood flow; diabetic retinopathy; microthrombosis; aspirin; clopidogrel
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy | interventions — Aspirin; Clopidogrel

INTERVENTIONS:
Drug: aspirin
Drug: clopidogrel

SUMMARY:
The project aims to find mechanisms for the abnormal retinal blood flow that in diabetic patients often precedes any evidence of clinical retinopathy and may contribute to the development of retinopathy.

Specifically, the projects tests the hypothesis that reduced retinal blood flow found in young patients with type 1 diabetes reflects increased resistance in the small vessels of the retina caused by the formation of small blood clots, called microthrombi; and that antiplatelet agents normalize the reduced retinal blood flow.

DETAILED DESCRIPTION:
The ultimate goal of this research is to contribute to the development of strategies to prevent diabetic retinopathy. This project will test the hypothesis that antiplatelet agents normalize the reduced blood flow observed early in the course of type 1 diabetes. If the hypothesis is proven correct, the results will indicate that the formation of small blood clots (microthrombi) occurs early in diabetic retinal vessels. In turn, because microthrombosis could readily account for the occlusive microangiopathy that causes the sight-threatening stages of diabetic retinopathy, the results will propose the desirability of antiplatelet therapy for the prevention of diabetic retinopathy.

We have three specific aims:

1. To confirm that, under basal conditions, retinal blood flow measured with the laser Doppler method in a group of type 1 diabetic patients with no or minimal retinopathy differs from the flow measured in age- and sex-matched nondiabetic control subjects;
2. To determine whether the response of retinal blood flow to low-dose aspirin (81 mg/day) administered for 2 months versus placebo, differs between type 1 diabetic patients with no or minimal retinopathy and age- and sex-matched nondiabetic control subjects;
3. To determine whether in type 1 diabetic patients with no or minimal retinopathy the response of retinal blood flow to low-dose aspirin differs from the response to clopidogrel, a drug that interferes with platelet function downstream of the site of aspirin action.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years,
* type 1 diabetes duration 1-15 years,
* absent or minimal retinopathy (EDTRS 20).
* Age- and gender-matched healthy controls

Exclusion Criteria:

* smoking,
* systemic diseases other than diabetes,
* retinal diseases other than diabetic retinopathy,
* pregnancy,
* bleeding disorders,
* aspirin allergy,
* use of anti-platelet agents,
* non-steroidal anti-inflammatory agents,
* angiotensin converting enzyme inhibitors,
* angiotensin receptor antagonists,
* Vitamin E in large doses.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2003-06; Study Completion 2006-03

PRIMARY OUTCOMES:
Retinal blood flow

SECONDARY OUTCOMES:
Retinal arterial blood speed
Retinal arterial diameter

CONTACTS AND LOCATIONS:
Overall Officials: Mara Lorenzi, MD, Principal Investigator — Schepens Eye Research Institute
Locations (1):
- Schepens Eye Research Institute, Boston, Massachusetts, United States